CLINICAL TRIAL: NCT06124807
Title: A Phase 2, Parallel-Group, Double-Blind, 4-Arm Study to Investigate Weight Management With LY3305677 Compared With Placebo and in Adult Participants With Obesity or Overweight
Brief Title: A Study of LY3305677 Compared With Placebo in Adult Participants With Obesity or Overweight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18661; W8M-MC-OXA1 (Other: ISA Number); CWMM Master Protocol (Other: Eli Lilly and Company); 2022-502816-35-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Overweight and Obesity
Keywords: Incretins; Weight Loss; Overnutrition
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Overnutrition | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3305677 Dose 1 (Experimental): Participants will receive LY3305677 subcutaneously (SC).
  Interventions: Drug: LY3305677
- LY3305677 Dose 2 (Experimental): Participants will receive LY3305677 SC.
  Interventions: Drug: LY3305677
- LY3305677 Dose 3 (Experimental): Participants will receive LY3305677 SC.
  Interventions: Drug: LY3305677
- Placebo (Placebo Comparator): Participants will receive LY3305677 matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3305677 — Administered SC
  Arms: LY3305677 Dose 1; LY3305677 Dose 2; LY3305677 Dose 3
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study, performed under a master protocol W8M-MC-CWMM (NCT06143956), is to investigate weight management efficacy and safety with LY3305677 compared with placebo and in adult participants with obesity or overweight. The study will last about 62 weeks.

ELIGIBILITY:
Inclusion Criteria:

W8M-MC-OXA1:

* Are males and females who agree to abide by the reproductive and contraceptive requirements

W8M-MC-CWMM:

* Have a BMI ≥27 kilograms per square meter (kg/m²)

Exclusion Criteria:

W8M-MC-OXA1:

* Have any prior diagnosis of diabetes mellitus, that is type 2 diabetes mellitus (T2DM), or rare forms of diabetes mellitus, except gestational diabetes.
* Have any of the following cardiovascular conditions within 6 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure (CHF).
* Have a history of acute or chronic pancreatitis.

  * Have a history of New York Heart Association (NYHA) Functional Classification I-IV CHF.
  * Participants with hypertension who do not have well-controlled blood pressure (BP) (>140/90 mmHg), regardless of antihypertensive treatment. Participants receiving treatment for hypertension should be on a stable antihypertensive regimen for at least 3 months prior to screening.

Note: If the investigator anticipates a need to add antihypertensive medication during the study, the participant should not be included in the ambulatory blood pressure monitoring (ABPM) procedures.

CWMM:

* Have a prior or planned surgical treatment for obesity, except prior liposuction or abdominoplasty, if performed >1 year prior to screening.
* Have type 1 diabetes mellitus, latent autoimmune diabetes in adults, or history of ketoacidosis or hyperosmolar coma.
* Have poorly controlled hypertension.
* Have signs and symptoms of any liver disease other than nonalcoholic fatty liver disease.
* Have a history of symptomatic gallbladder disease within the past 2 years.
* Have a lifetime history of suicide attempts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline to Week 32

SECONDARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 48
Change from Baseline in Body Weight | Baseline, Week 32
Change from Baseline in Body Weight | Baseline, Week 48
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Baseline to Week 32
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Baseline to Week 48
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Baseline to Week 32
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Baseline to Week 48
Change from Baseline in Body Mass Index (BMI) | Baseline to Week 32
Change from Baseline in BMI | Baseline to Week 48
Number of Participants with Treatment Emergent Drug Antibodies (TE-ADAs) | Baseline to Week 56
Pharmacokinetics (PK): Area Under the Curve (AUC) of LY3305677 | Baseline to Week 56
PK: Maximum Concentration (Cmax) of LY3305677 | Baseline to Week 56
Absolute Change from Baseline in Liver Fat Content (LFC) by Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) in Participants with Baseline LFC≥5% and Baseline LFC≥10% | Baseline to Week 32
Percent Change from Baseline in Liver Fat Content by MRI-PDFF in Participants with Baseline LFC≥5% and Baseline LFC≥10% | Baseline to Week 32
Absolute Change from Baseline in Liver Fat Content by MRI-PDFF in Participants with Baseline LFC ≥5% and Baseline LFC≥10% | Baseline to Week 48
Percent Change from Baseline in Liver Fat Content by MRI-PDFF in Participants with Baseline LFC ≥5% and Baseline LFC≥10% | Baseline, Week 48
Percentage of Participants Who Achieve ≥30% Relative Reduction in LFC | Baseline to Week 32
Percentage of Participants Who Achieve >30% Relative Reduction in LFC | Baseline to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- United States (29):
  - The Institute for Liver Health II dba Arizona Clinical Trials - Mesa, Chandler, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health-Tucson, Tucson, Arizona
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Knownwell, Needham, Massachusetts
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - North Suffolk Neurology, Port Jefferson Station, New York
  - Lucas Research, Inc., New Bern, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Quality Medical Research, Nashville, Tennessee
  - IMA Clinical Research Austin, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Tekton Research - Fredericksburg Road, San Antonio, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Plan Description:
  Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of LY3305677 Compared With Placebo in Adult Participants With Obesity or Overweight — https://trials.lilly.com/en-US/trial/434975